CLINICAL TRIAL: NCT05495672
Title: Circulating Tumor DNA Guided Therapeutic Strategies for Colorectal Cancer Patients With Small Pulmonary Nodules Suspected to be Metastases: an Open-Label, Prospective, Phase II Cohort Study
Brief Title: Circulating Tumor DNA Guided Therapeutic Strategies for CRC Patients With Small Pulmonary Nodules
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Junjie Peng (Other)
Collaborators: Shanghai OrigiMed Co., Ltd. (Unknown)
Responsible Party: Sponsor-Investigator, Junjie Peng, MD, PhD, Fudan University
Organization: Fudan University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ctDNA-nedCRC-lung
Record Dates: First submitted 2022-07-26; First posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Advanced Colorectal Cancer; Circulating Tumor DNA
Keywords: advanced colorectal cancer; lung metastasis; circulating tumor DNA

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1-Arm A: the largest pulmonary nodule is less than or equal to 1 cm, ctDNA positive (Experimental): ctDNA is detected before curative treatment. Subjects with ctDNA positive before treatment will receive curative treatments for pulmonary nodules such as surgery, radio frequency ablation or stereotactic body radiotherapy. ctDNA will be detected after curative treatment and then every three months until progression or 2 years. At the same time, routine post treatment follow-up will be performed.
  Interventions: Procedure: Local treatment
- Cohort 1-Arm B: the largest pulmonary nodule is less than or equal to 1 cm, ctDNA negative (No Intervention): Subjects with ctDNA negative will undergo routine follow-up. ctDNA will be detected every three months until progression or 2 years.
- Cohort 2-Arm C: the largest pulmonary nodule is between 1 cm to 2 cm, ctDNA positive (Experimental): ctDNA is detected before curative treatment. Subjects with ctDNA positive before treatment will receive curative treatments for pulmonary nodules such as surgery, radio frequency ablation or stereotactic body radiotherapy.
  ctDNA is rechecked following treatment. Subjects with ctDNA positive after treatment will receive chemotherapy. Subjects with ctDNA negative after curative treatment will undergo routine follow-up.
  After treatment, ctDNA will be detected every three months until progression or 2 years. At the same time, routine post treatment follow-up will be performed.
  Interventions: Procedure: Local treatment
- Cohort 2-Arm D: the largest pulmonary nodule is between 1 cm to 2 cm, ctDNA negative (No Intervention): Subjects with ctDNA negative will undergo routine follow-up. ctDNA will be detected every three months until progression or 2 years.

INTERVENTIONS:
Procedure: Local treatment — Radical surgical resection, local radiotherapy, radiofrequency ablation (RFA) or interventional therapy (absolute alcohol or cryotherapy).
  The equipment used for RFA of lung lesions consisted of the radiofrequency generator (CelonLab POWER), cold circulation pump (Celon Aquaflow Ⅲ), radiofrequency needle electrode (Celon proSurge: T20, T30 and T40 is an electrode length of 20, 30 and 40 mm respectively, and maximum output power of 20, 30 and 40 W; Olympus Surgical Technologies Europe, Hamburg, Germany).
  Arms: Cohort 1-Arm A: the largest pulmonary nodule is less than or equal to 1 cm, ctDNA positive; Cohort 2-Arm C: the largest pulmonary nodule is between 1 cm to 2 cm, ctDNA positive

SUMMARY:
The clinical diagnosis and treatment of small pulmonary nodules (suspected to be lung metastases) in advanced colorectal cancer patients remain controversy. Previous studies have shown that tumor-informed circulating tumor DNA (ctDNA) blood testing can sensitively detect residual cancer. Postoperative ctDNA in colorectal cancer patients is a valuable biomarker to identify minimal residual disease (MRD) after radical resection, which is possibly useful in redefining the risk group of patients and guiding postoperative treatment. This study aimed to explore the clinical value of therapeutic strategies based on tumor-informed ctDNA test in advanved colorectal cancer patients with small pulmonary nodules.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤80 years old, regardless of gender;
2. Pathologically confirmed as adenocarcinoma of advanced colorectal cancer;
3. Lung lesions only, which was considered as metastatic by imaging consultation, and clinically diagnosed as lung metastasis of colorectal cancer;
4. Multiple lung lesions are allowed, but the maximum lesion diameter should be less than or equal to 2 cm;
5. For lesions larger than 1 cm, local treatment is planned, such as radical surgical resection or local radiotherapy, radio frequency ablation or interventional therapy (absolute alcohol treatment or cryotherapy);
6. Eastern Cooperative Oncology Group (ECOG) score 1 ~ 2;
7. The subjects (or their legal representative / Guardian) must sign the informed consent form, indicating that they understand the purpose of the study, understand the necessary procedures of the study, and are willing to participate in the study;
8. Surgical specimens or puncture specimens containing tumor tissue are available;
9. 20 mL of peripheral blood are available (10 mL per tube, two tubes in total);
10. Agreed to follow up for at least 2 years.

Exclusion Criteria:

1. The pathology was not confirmed by enteroscopic biopsy or biopsy of metastatic lesions;
2. Patients with stage I-III colorectal cancer;
3. Primary lung cancer, GGO, tuberculosis and other non metastatic conditions were excluded after diagnosis by imaging consultation;
4. Presence of metastasis other than lung;
5. Insufficient organ function, such as severe abnormal hemogram, abnormal liver and kidney function;
6. Any signs of severe or uncontrolled systemic diseases that the researcher believes may have a significant patient risk/benefit balance, including uncontrolled hypertension, severe infection, hepatitis B, hepatitis C and human immunodeficiency virus;
7. History of alcoholism or drug abuse;
8. Pregnant or lactating patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) in advanced colorectal cancer patients with metastatic small pulmonary nodules under ctDNA guided therapeutic strategies | From date of treatment until the date of first documented progression or date of death from any cause, assessed up to 36 months.

SECONDARY OUTCOMES:
ctDNA positive rate in colorectal cancer patients with metastatic small pulmonary nodules | 4 weeks
ctDNA positive prediction rate (Consistent with histopathological result as the standard for comparison) | 8 weeks
The ctDNA clearance rate after local treatment | 8 weeks
The ctDNA clearance rate after chemotherapy in patients achieving NED (Cohort 2) | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No